CLINICAL TRIAL: NCT03059030
Title: Yttrium-90 Radioembolization for Cirrhosis-Associated Thrombocytopenia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Northwestern University (Other)
Collaborators: BTG International Inc. (Other)
Responsible Party: Principal Investigator, Riad Salem, Chief, Vascular and Interventional Radiology, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 00203772
Record Dates: First submitted 2017-02-08; First posted 2017-02-23 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Thrombocytopenia; Cirrhosis
Keywords: Thrombocytopenia; cirrhosis; Therasphere®; Y90; Radioembolization
MeSH Terms: conditions — Thrombocytopenia; Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Subjects with thrombocytopenia secondary to cirrhosis (Experimental): Evaluate the safety and efficacy of 90Y radioembolization for the management of thrombocytopenia.
  Interventions: Device: TheraSphere® Yttrium-90 Glass Microspheres, BTG International Inc.

INTERVENTIONS:
Device: TheraSphere® Yttrium-90 Glass Microspheres, BTG International Inc. — The Interventional Radiologists will inject a dose of Yttrium 90 into your spleen through a small catheter placed in your femoral artery.The entire treatment visit is an outpatient procedure. You will only be admitted to the hospital if the physician deems it necessary due to any symptoms you may experience after the treatment is given. This visit may take 6 to 8 hours.

SUMMARY:
Evaluate the safety and efficacy of Yttrium-90 (90Y) radioembolization for the management of thrombocytopenia.

DETAILED DESCRIPTION:
This protocol will provide access to TheraSphere® treatment for patients who have refractory thrombocytopenia secondary to cirrhosis. This protocol will utilize splenic artery-directed TheraSphere® treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years of age or older, of any ethnic or racial group.
* Diagnosis of cirrhosis or portal hypertension with a serum platelet count less than or equal to 80 × 109/L. [Rationale: platelet count <100 × 109/L triples the rate of liver-related adverse events (3) and worsens postoperative survival in the setting of hepatocellular carcinoma (HCC) (4). Initial platelet count of 80 × 109/L can allow the majority of patients who successfully respond to 90Y-RE (clinical endpoint of 50% platelet count increase) to exceed the 100 × 109/L threshold.]

Cirrhosis is defined by one of three criteria:

* Liver Biopsy/histology consistent with cirrhotic architectural liver changes
* Portal hypertension (Hepatic venous pressure gradient ≥10 mm Hg)
* Evidence of esophageal and/or gastric varices
* Patients must have evidence of splenomegaly as determined by screening cross-sectional imaging.
* No evidence of myelosuppression (e.g. lymphopenia) as evidenced by normal hematology values at Screening
* Adequate baseline organ function(with the exception of cirrhosis) as evidenced by normal BUN/Cr and electrolytes on screening chemistry.
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0-2
* Patient has a life expectancy of greater than 6 months without intervention.
* Patient is willing to participate in the study and has signed the study informed consent.
* Women of childbearing potential must have a negative serum pregnancy test within 28 days prior to screening and must not be breastfeeding.

Exclusion Criteria:

* Patients with serum platelet count less than 10 × 109/L.
* History of bleeding disorder attributed to another cause other than cirrhosis (e.g. Von Willebrand disease)
* Declines or unable to provide informed consent
* History of prior partial splenic embolization (PSE) or splenectomy
* Use of any medication known to increase platelet count 1 month prior to Baseline.
* History of allergy or sensitivity to TheraSphere® or its components.
* History of severe peripheral allergy or intolerance to contrast agents, narcotics, sedatives or atropine that cannot be managed medically
* Contraindications to angiography and selective visceral catheterization such as bleeding, diathesis or coagulopathy that is not correctable by usual therapy or hemostatic agents (e.g. closure device)
* Previous randomization in a trial using 90Y RE
* Patient must not have participated or enrolled in a clinical trial with an investigational device / therapy within 30 days prior to randomization
* Any serious medical condition likely to impede successful completion of the study, such as certain mental disorders, cardiac arrhythmias, and uncontrolled congestive heart failure or respiratory disease.
* Patients actively on chemotherapy.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2017-03-16 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Riad Salem, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University/Northwestern Memorial Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Subjects With Thrombocytopenia Secondary to Cirrhosis: Evaluate the safety and efficacy of 90Y radioembolization for the management of thrombocytopenia.
  TheraSphere® Yttrium-90 Glass Microspheres, BTG International Inc.: The Interventional Radiologists will inject a dose of Yttrium 90 into your spleen through a small catheter placed in your femoral artery.
Period: Overall Study
Arm/Group | Subjects With Thrombocytopenia Secondary to Cirrhosis
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: To evaluate the safety and efficacy of yttrium-90 transarterial radioembolization (90Y TARE) for cirrhosis-associated thrombocytopenia for the purpose of decreasing splenic size and increasing platelet counts.
Arm/Group | Subjects With Thrombocytopenia Secondary to Cirrhosis
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] | 61 [47 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: The Primary Objective of This Pilot Study is to Evaluate the Safety of 90Y TARE for the Treatment of Thrombocytopenia in the Setting of Cirrhosis. Evaluation of Overall AE Reporting in All Categories.
Description: The number and the severity of ALL adverse events will be recorded to evaluate safety. Events will be reported by subjects at follow up visits.
  Scale: Common Terminology Criteria for Adverse Events (CTCAE) CT CAE v 4.0.3 Grades range from 1-5 with 5 being the worst (Death), descriptions of each grade for specific AE's are available here: https://evs.nci.nih.gov/ftp1/CTCAE/CTCAE_4.03/CTCAE_4.03_2010-06-14_QuickReference_8.5x11.pdf Total AE's of different types are collected and for each grade are reported as a group
Time Frame: 6 months
Population: All subjects enrolled received treatment per protocol.
Measure: Number; unit: events
Groups:
- Subjects With Thrombocytopenia Secondary to Cirrhosis: There is only one arm of the study where patients received treatment.
Arm/Group | Subjects With Thrombocytopenia Secondary to Cirrhosis
Number analyzed (Participants) | 7
events
  Grade 1 AE | 49
  Grade 2 AE | 34
  Grade 3 AE | 28
  Grade 4 AE | 15
  Grade 5 AE | 0

2. Primary Outcome: Safety of 90Y RE for the Treatment of Thrombocytopenia in the Setting of Cirrhosis. Reporting of Splenic Abscess.
Description: The number and the severity of adverse events related to splenic abscess will be recorded to evaluate safety. Events will be reported by subjects at follow up visits.
  Scale: Common Terminology Criteria for Adverse Events (CTCAE) CT CAE v 4.0.3 Grades range from 1-5 with 5 being the worst (Death), Grade 1 (Mild):Small abscess with minimal symptoms, often not requiring intervention.
  Grade 2 (Moderate):Larger abscess causing moderate symptoms, may require antibiotics or drainage procedures.
  Grade 3 (Severe):Large abscess with significant symptoms, potentially causing systemic effects, requiring hospitalization and aggressive management.
  Grade 4 (Life-threatening):Abscess with immediate life-threatening complications, requiring urgent intervention.
  Grade 5 Death
Time Frame: 6 months
Population: All subjects treated on study.
Measure: Number; unit: events
Arm/Group | Subjects With Thrombocytopenia Secondary to Cirrhosis
Number analyzed (Participants) | 7
events
  Grade 1 | 0
  Grade 2 | 0
  Grade 3 | 0
  Grade 4 | 0
  Grade 5 | 0

3. Primary Outcome: Safety of 90Y RE for the Treatment of Thrombocytopenia in the Setting of Cirrhosis. AE's Related to Infection.
Description: The number and the severity of adverse events related to infection will be recorded to evaluate safety. Events will be reported by subjects at follow up visits.
  Common Terminology Criteria for Adverse Events (CTCAE) CT CAE v 4.0.3, Grades range from 1-5 with 5 being the worst (Death) Grade 1 (Mild): Asymptomatic or mild symptoms, only requiring clinical observation, no intervention needed.
  Grade 2 (Moderate): Symptoms limiting some daily activities, minimal intervention may be required.
  Grade 3 (Severe): Symptoms significantly impacting self-care, requiring hospitalization or prolonged stay.
  Grade 4 (Life-threatening): Urgent intervention needed due to life-threatening complications.
  Grade 5 (Death): Death directly related to the infection.
Time Frame: 6 months
Population: 3 subjects reported infections these were unrelated to treatment on study. Pneumonia grade 3, lung infection grade 3, vaginal infection grade 2. All resolved before the study was completed.
Measure: Number; unit: events
Arm/Group | Subjects With Thrombocytopenia Secondary to Cirrhosis
Number analyzed (Participants) | 7
events
  Grade 1 | 0
  Grade 2 | 1
  Grade 3 | 2
  Grade 4 | 0
  Grade 5 | 0

4. Primary Outcome: Asses the Need for Technetium Albumin Aggregated (TC-MAA 99m) Injection to Determine Shunting Prior to Y90 Administration
Description: MAA injection will be done and nuclear medicine PET scan to evaluate shunting and evaluated for the first 4 patients. If shunt is <5% subsequently enrolled patients will not undergo MAA, if shunt is >5% all subsequent patients will undergo MAA. This will be evaluated post MAA injection before Y90 treatment.
Time Frame: 6 months
Population: All four patients that received Tc-MAA to determine shunting prior to Y90 RE had a lung shunt fraction <5%. Given this finding no subsequent patients needed MAA or lung shunt study performed.
Measure: Number; unit: participants
Arm/Group | Subjects With Thrombocytopenia Secondary to Cirrhosis
Number analyzed (Participants) | 4
participants | 0

5. Secondary Outcome: Achieve a 50% Increase in Platelet Count Six Months After Therapy.
Description: Complete Blood Count with platelets will be drawn at baseline, treatment, 2, 4, 6, 8 weeks and 3, 4, 5, 6 months post treatment. Comparison made with screening platelet count and 6 month follow up visit platelet count.
Time Frame: 6 months
Population: The 7 participating subjects had platelets drawn 6 months post procedure.
Measure: Number; unit: participants
Arm/Group | Subjects With Thrombocytopenia Secondary to Cirrhosis
Number analyzed (Participants) | 7
participants
  Achieved 50% increase in 6 months | 0
  Did not achieve 50% increase in 6 months | 7

6. Secondary Outcome: Achieve 20% Decrease in Functional Splenic Volume Six Months After Treatment
Description: Assessed via cross sectional CT or MR of the abdomen at screening and at 4 weeks, 3 months, and 6 months post treatment. Comparison made with screening CT or MR and 6 month follow up imaging.
Time Frame: 6 months
Population: All subjects had a CT or MR at screening, 1 month, 3 months, and 6moths timepoints. Splenic volumes were reported at all time points.
Measure: Number; unit: participants
Arm/Group | Subjects With Thrombocytopenia Secondary to Cirrhosis
Number analyzed (Participants) | 7
participants
  Achieved 20% decrease in volume | 1
  Did not achieve 20% decrease in volume | 6

7. Secondary Outcome: Evaluate Length of Hospital Stay After Procedure
Description: Determine the average length of stay in the hospital in days after treatment.
Time Frame: 6 months
Population: no subjects were admitted after their procedure so there are 0 days hospitalized to report or analyze.
Arm/Group | Subjects With Thrombocytopenia Secondary to Cirrhosis
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse events were collected at all follow up visits: 2 weeks, 1 month, 6 weeks, 2, 3, 4, 5, and 6 months post procedure.
Groups:
- Subjects With Thrombocytopenia Secondary to Cirrhosis: Evaluate the safety and efficacy of 90Y radioembolization for the management of thrombocytopenia. TheraSphere® Yttrium-90 Glass Microspheres, BTG International Inc.: The Interventional Radiologists will inject a dose of Yttrium 90 into your spleen through a small catheter placed in your femoral artery. There was only one arm of this study and all subjects were treated.
  No subjects had severe adverse events and none died during the duration of the study. All adverse events reported at follow up visits were reported.
Arm/Group | Subjects With Thrombocytopenia Secondary to Cirrhosis
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 7/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Subjects With Thrombocytopenia Secondary to Cirrhosis (N=7)
White Blood Cell Count Decreased (Blood and lymphatic system disorders) | 6 (7)
Lymphocyte Count Decreased (Blood and lymphatic system disorders) | 7 (7)
Anemia (Blood and lymphatic system disorders) | 5 (6)
Neutrophil count decreased (Blood and lymphatic system disorders) | 5 (5)
Alkaline Phosphatase Increased (Hepatobiliary disorders) | 2 (2)
Ascites (Hepatobiliary disorders) | 3 (3)
Fatigue (General disorders) | 5 (6)
Anorexia (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 3 (3)
Presyncope (General disorders) | 1 (1)
Chest Pain (Cardiac disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 2 (2)
Pain in extremity (General disorders) | 1 (1)
Limb Edema (Blood and lymphatic system disorders) | 2 (2)
Upper GI Hemorrhage (Gastrointestinal disorders) | 1 (1)
Acute Kidney injury (Renal and urinary disorders) | 1 (1)
Hyperkalemia (Endocrine disorders) | 1 (1)
Hypokalemia (Endocrine disorders) | 2 (3)
Hypocalcemia (Endocrine disorders) | 3 (4)
Hypoalbuminemia (Hepatobiliary disorders) | 4 (4)
Hyponatremia (Endocrine disorders) | 4 (4)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 2 (2)
Vaginal Infection (Reproductive system and breast disorders) | 1 (1)
Lower GI Hemorrhage (Gastrointestinal disorders) | 1 (1)
Knee Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cholesterol High (Blood and lymphatic system disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 3 (5)
Hiccupping (Gastrointestinal disorders) | 1 (1)
Decreased Platelet Count (Blood and lymphatic system disorders) | 3 (3)
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Increased Cardiac Troponin I (Cardiac disorders) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Bruising (General disorders) | 1 (1)
Right Ventricular Dysfunction (Cardiac disorders) | 1 (1)
Hot Flashes (General disorders) | 1 (1)
Chronic Kidney Disease (Renal and urinary disorders) | 1 (1)
Hernia Pain (Gastrointestinal disorders) | 1 (1)
Genital Edema (Blood and lymphatic system disorders) | 1 (1)
Scrotal Pain (Reproductive system and breast disorders) | 1 (1)
Wound Dehiscence (General disorders) | 1 (1)
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 (1)
Lung Infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Benign neoplasm -Antral polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Edema Face (Blood and lymphatic system disorders) | 1 (1)
Blood Bilirubin increased (Hepatobiliary disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Chills (General disorders) | 2 (2)
INR Increased (Blood and lymphatic system disorders) | 1 (1)
Hypertension (Cardiac disorders) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1)
Insomnia (General disorders) | 1 (1)
Pelvic Pain (General disorders) | 1 (1)
Weight Loss (General disorders) | 1 (1)
Worsening GI Reflux (Gastrointestinal disorders) | 1 (2)
Aspartate Aminotransferase Increased (Blood and lymphatic system disorders) | 1 (1)
Dizziness (General disorders) | 1 (1)
Increased Creatnine (Renal and urinary disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Skin disorder Atypical nevi abdomen (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperglycemia (Endocrine disorders) | 1 (2)

LIMITATIONS AND CAVEATS:
Enrollment in the clinical trial did not reach the target number of subjects needed to achieve target power and was insufficient to produce statistically reliable results. There were too few eligible candidates or willing participants over several years even with several clinics and a multidisciplinary team reviewing potential candidates. The trial was terminated for low enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-07): https://cdn.clinicaltrials.gov/large-docs/30/NCT03059030/Prot_SAP_000.pdf